CLINICAL TRIAL: NCT07361276
Title: Clinical Landscape of Epidemiology and Assessment of Results in Hypertension
Brief Title: Observational Study That Will Evaluate Treatment Patterns in the Management of Hypertension in Various Scenarios in the Public Primary Care System
Acronym: CLEAR-HTN
Status: Not yet recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D6970R00015
Record Dates: First submitted 2026-01-14; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-09

CONDITIONS: Hypertension
Keywords: Blood Pressure, High
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective observational cohort study based on secondary use of routinely collected electronic health data. The design was selected to enable population-level characterisation of treatment patterns and clinical inertia (both diagnostic and therapeutic) in the management of hypertension across diverse settings in Brazil's public primary care system (SUS).

DETAILED DESCRIPTION:
This is a retrospective observational cohort study based on secondary use of routinely collected electronic health data. The design was selected to enable population-level characterisation of treatment patterns and clinical inertia (both diagnostic and therapeutic) in the management of hypertension across diverse settings in Brazil's public primary care system (SUS).

The retrospective cohort design allows for efficient use of existing clinical data to evaluate real-world practice against national guideline recommendations. The primary outcomes relate to treatment decisions and delays rather than interventional effects; therefore, an observational design is methodologically appropriate and ethically preferable.

The study will be conducted across 05 Brazilian municipalities participating in the epHealth Primary Care Solutions platform. These municipalities span multiple regions and reflect heterogeneity in socio-demographic context, healthcare infrastructure, and epidemiological profiles.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at the time of Hypertension diagnosis
* Hypertension diagnosis as retrieved from registered ICD codes or CIAP Codes (primary care codes) in the EMR , OR At least two blood pressure measurements ≥140/90 mmHg during the study period. The blood measurements should be consecutive and obtained within a 30 days period.
* Continuous follow-up in the same municipality for at least 6 months after index measurement.
* Availability of structured EMR data including clinical encounters, diagnoses, and prescriptions

Exclusion Criteria:

- Patients with incomplete data or not traceable in the registration systems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults registered in the e-SUS PEC system who had encounters with primary healthcare services within the study period and had blood pressure measurements recorded. We will assess data from the entire population of approximately 05 muncipalities (comprising between 100.000 and 250.000 inhabitants). The municipalities will be seleceted from a pre-screened list of 20 cities located within all Brazilian regions.
Sampling Method: Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Uncontrolled blood pressure | through study completion, an average of 1 year
  Proportion of patients with uncontrolled blood pressure (BP ≥ 140/90 mmHg) who did not receive treatment intensification within 3 months of a recorded elevated BP.

SECONDARY OUTCOMES:
Antihypertensive treatment | through study completion, an average of 1 year
  Proportions receiving monotherapy vs. combination therapy; distribution by pharmacologic class.
Risk stratification | through study completion, an average of 1 year
  Likelihood of treatment escalation stratified by low/moderate vs. high/very high CV risk.

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal
  Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org